CLINICAL TRIAL: NCT02997332
Title: Phase I Trial Evaluating the Safety of Durvalumab in Combination With Docetaxel, Cisplatin and 5-FU in Induction for Locally Advanced Head and Neck Squamous Cell Carcinoma
Brief Title: Durvalumab in Combination With Docetaxel, Cisplatin and 5-FU for Locally Advanced Head and Neck Squamous Cell Carcinoma
Acronym: MEDINDUCTION
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-004146-25; 2015/2316 (Other: CSET number)
Record Dates: First submitted 2016-12-13; First posted 2016-12-20 (Estimated); Last update posted 2019-01-03 (Actual); Status verified 2019-01

CONDITIONS: Head and Neck Cancers
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — durvalumab; Docetaxel; Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with squamous cell carcinoma of the oral cavity, (Experimental): The aim is to evaluate safety, PK and pharmacodynamics of durvalumab in adult patients with squamous cell carcinoma of the oral cavity, oropharynx, larynx or hypopharynx previously untreated, with indication of induction chemotherapy.
  Interventions: Drug: Durvalumab; Drug: Docetaxel; Drug: Cisplatin; Drug: 5 Fluorouracil

INTERVENTIONS:
Drug: Durvalumab — Durvalumab will be administered every 3 weeks for 3 injections at week 1, 4, 7. Dose levels: the durvalumab first dose level is 1120 mg Q3W, and the dose level -1 is 750 mg Q3W.
Drug: Docetaxel — Docetaxel 75mg/m² on D2, IV in 1 hour
Drug: Cisplatin — Cisplatin 75mg/m² on D2, IV in 3 hours
Drug: 5 Fluorouracil — 5 Fluorouracil 750mg/m²/day on D2, D3, D4, D5, D6 IV in 24 hours

SUMMARY:
The prognosis of patients with locally advanced SCCHN is poor. Results of recent randomized trials evaluating induction chemotherapy by docetaxel, cisplatin, 5 fluorouracil are conflicting, and benefit on overall survival is uncertain. Improve efficacy of induction chemotherapy is important without increase toxicities. Durvalumab is a promising agent in SSCHN. The safety of combination of docetaxel, cisplatin, 5 fluorouracil with durvalumab is unknown.

The aim of the study is to evaluate the feasibility and the safety of the association of DCF (standard regimen for induction in SSCCHN) and durvalumab. The safety profile of DCF and durvalumab are different, so the expected toxicities should not be additive. The addition of durvalumab to DCF could improve the efficacy of induction chemotherapy and the prognostic of patients with SSCCHN.

Concerning the translational research, the aim will be to explore the relationships between immune capacity, specificity, activation state and clinical outcome to help elucidate the determinants of response to immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years and < 75 years
2. Histologically or cytologically confirmed squamous cell carcinoma of the oral cavity, oropharynx, larynx or hypopharynx, previously untreated, amenable to induction chemotherapy according to the investigator. Patients with a diagnosis of SCCHN of occult primary could be enrolled.
3. Absence of metastases determined by CT scan or PET scan
4. ECOG performance status < 1
5. Subjects must have at least 1 measurable lesion per RECIST v1.1 guidelines
6. Adequate organ and marrow function as defined below:

   * Hemoglobin ≥ 9,0 g/dL
   * Absolute neutrophil count (ANC) ≥ 1,500/mm3
   * Platelet count ≥ 100,000/mm3
   * AST and ALT ≤ 2.5 × institutional upper limit of normal (ULN);
   * Total bilirubin ≤ 1.5 × ULN;
   * Creatinine clearance > 60 mL/min as determined by the Cockcroft-Gault equation (Cockcroft and Gault, 1976) or by 24-hour urine collection for determination of creatinine clearance
7. Negative serology for hepatitis B and C
8. Availability of a recent formalin-fixed tumour tissue (< 3 months) to determine HPV status and for translational research (IHC)

   a. All patients without available tumour tissue will undergo a panendoscopy with biopsies.
9. Women of childbearing potential must have a negative serum β-HCG pregnancy test within 7 days prior to the administration of the first study treatment and/or urine pregnancy 48 hours prior to the administration of the first study treatment. Both sexually active women of childbearing potential and males (and their female partners) patients must agree to use two methods of effective contraception, one of them being a barrier method, or to abstain from sexual activity during the study and for at least 6 months after last dose of study drugs.
10. Patients must be willing and able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures
11. Patients must be affiliated to a Social Security System or beneficiary of the same
12. Patient information and written informed consent form signed

Exclusion Criteria:

1. Primary site of head and neck carcinoma in nasopharynx, or skin
2. Patients receiving other anti-cancer medication such as, chemotherapy, immunotherapy, biologic therapy, targeted therapy, monoclonal antibodies, hormonal therapy (other than leuprolide or other GnRH agonists) or other investigational agent within 30 days prior to the first dose of study drug and while on study treatment.
3. Patients receiving other anti-cancer non-drug therapies: radiation, or tumor embolization within 30 days prior to the first dose of study drug and while on study treatment.
4. No relevant toxicities (>grade 1 CTCAE) due to prior medical treatment at time of study entry
5. Participation in another clinical study with an investigational product during the last 30 days
6. Patient with dihydropyrimidine dehydrogenase (DPD) deficiency
7. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, active peptic ulcer disease or gastritis, active bleeding diatheses. Or patient under guardianship or deprived of his liberty by a judicial or administrative decision or any condition (e.g psychiatric illness/social/familial/geographical condition) that would limit compliance with study requirement or compromise the ability of the subject to give written informed consent
8. Patient with active cardiac disease or with a history of cardiac dysfunction any of the following:

   * Left Ventricular Ejection Fraction (LVEF) < 50% as determined by Multiple Gated acquisition (MUGA) scan or echocardiogram (ECHO),
   * Mean QT interval corrected for heart rate (QTc) ≥ 470 msec calculated from 3 electrocardiograms (ECGs) performed at screening, using Fredericia's correction (QTcF),
   * Myocardial infarction within the last 6 months, documented by persistent elevated cardiac enzymes or persistent regional wall abnormalities on assessment of LVEF function,
   * Unstable angina pectoris
   * Uncontrolled hypertension
   * History of documented congestive heart failure (New York Heart Association functional classification III-IV), or Uncontrolled symptomatic congestive heart failure
   * Documented cardiomyopathy,
   * Other cardiac arrhythmia not controlled with medication.
9. Other invasive malignancy within 5 years except for noninvasive malignancies such as cervical carcinoma in situ, non-melanomatous carcinoma of the skin or ductal carcinoma in situ of the breast that has/have been surgically cured
10. Current or prior use of immunosuppressive medication within 28 days before the first dose of durvalumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone or an equivalent corticosteroid
11. Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving durvalumab
12. Active or prior documented autoimmune disease within the past 2 years NOTE: Subjects with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded
13. Active or prior documented inflammatory bowel disease (eg, Crohn's disease,ulcerative colitis)
14. History of primary immunodeficiency
15. History of allogenic organ transplant that requires use of immunosuppressives
16. Known history of previous clinical diagnosis of tuberculosis
17. Patients with a known HIV status
18. Pregnant or breast-feeding women
19. Any previous treatment with a PD1 or PD-L1 inhibitor, including durvalumab
20. History of hypersensitivity to durvalumab or any excipients or to other humanized mAbs
21. Any contraindication to the use of cisplatin, docetaxel and 5FU and/or known history of hypersensitivity to any of those drugs
22. Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2017-03-30 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase 2 dose (RP2D) | Up to 10 weeks
  To determine the recommended Phase 2 dose (RP2D) and schedule of durvalumab when administered with docetaxel, cisplatin and 5 Fluorouracil
Number of Dose Limiting Toxicity (DLT) | Up to 6 weeks
  To characterize the safety and tolerability profile of durvalumab when administered in combination with docetaxel, cisplatin and 5 Fluorouracil

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy, Villejuif, Val De Marne, France

IPD SHARING:
Plan to Share IPD: No